CLINICAL TRIAL: NCT04824183
Title: A Pilot Study on the Effect of Culturally-adapted Music Intervention on Preoperative Anxiety and Acute Postoperative Pain Among African Women Undergoing Mastectomy: A Randomised Controlled Trial
Brief Title: Music Intervention for Preoperative Anxiety and Acute Pain Among Mastectomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Yetunde Oluwafunmilayo TOLA, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021.127
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer; Mastectomy; Pain, Postoperative
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Single-blind multicenter randomised controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music intervention (Experimental): Music intervention that begins with patient education on WhatsApp will be delivered to participants 3 times within 48 hours before surgery followed by face-to-face monitoring of intervention usage.
  Interventions: Other: Music intervention
- Usual care (No Intervention): Participants in the control group will receive preoperative pain education via a one-on-one WhatsApp chat. The pain education will focus mainly on the type of pain to expect after surgery, how to report pain and how to request pain medication. MI will not be introduced to the participants in this group neither will there be any phone call for psychological support. Other preoperative care and postoperative care will be provided according to the hospital and ward practices.

INTERVENTIONS:
Other: Music intervention — Three WhatsApp sessions will be delivered before the surgery. In the first session, participants will describe their experience with the diagnosis of breast cancer and acceptance. In the second session, participants will be educated on anxiety before their surgery, how anxiety is being managed in the hospital and self-care strategies for anxiety like MI, how to report preoperative anxiety. The third session will include postoperative pain education. The pain education will include information about the type of pain to expect after surgery, medications, pain reporting and MI for pain management. Telephone session; on the day of surgery and at 24 and 48 hours after surgery, a reminder will be sent to the participants by WhatsApp group chat. Face-to-face; MI delivery will involve the delivery of the MP3 to participants and monitoring of their use for 30 minutes both on the day of surgery and 24 and 48 hours after surgery.
  Other Names: Hybrid-mode delivered music intervention
  Arms: Music intervention

SUMMARY:
Anxiety is a common thing that patients experience when they are preparing to have a surgery. When this anxiety is not properly treated, the patients tend to consume more drugs in the operating room and it also cause their pain to increase after surgery. Pain after surgery is common among patients who have just had surgery. The pain that women who have had mastectomy feels after surgery is usually treated using pain killers. Yet, the pain killers are not enough to reduce the pain or cause some unwanted outcomes for the patients. Therefore, supplementing pain killers with music therapy appears to be a good way to reduce the pain and the unwanted outcomes that may arise from taking too much pain killers.

This research is aimed to test how effective music that is selected by patients, considers their culture and psychological needs can be helpful in reducing anxiety before surgery and pain after surgery. Also its effect on blood pressure, breathing rate and pulse will be tested. The researcher also hope to know how satisfied patients who consent to participate in the study are with their pain management.

The study will be done in two Nigerian hospitals and will mainly include women who have cancer, are above the age of 18, scheduled to have mastectomy, can read or write English or Pidgin, without any mental health challenge and agrees to participate in the study.

This study hope to enrol up to 112 women and put them into two groups randomly, one group will receive the music intervention and the other group will receive the normal care provided by the hospital.

Participants in the music intervention group will be added to a WhatsApp group on the week of their surgery. The WhatsApp session will be three times within the week of the surgery and each session will be about 30 minutes long. This study will use a combination of very short videos and voice notes (3 minutes) as well as real time chats and pictures to enhance communication on the group chat. The researcher will initiate discussions about participant's experience with breast cancer diagnosis, teach them about anxiety before surgery and pain after surgery. Then, they will ask questions that will be answered and also choose their type of music and send it to the group. The songs will be downloaded into a device and given to them on the day of surgery. They will continue to listen to the music after their surgery for the next two days.

Before participants receive the music on the day of surgery, anxiety level and vital signs will be assessed. After the surgery, participant's pain level, vital signs and satisfaction with pain management before and after the intervention will be assessed. Those in the second group will receive a one-on-one chat with the researcher about pain after surgery.

For all the participants, the study will be completed two days after the surgery.

DETAILED DESCRIPTION:
Music intervention (MI) is considered useful for anxiety and pain management in various surgical populations. It is a mind-body therapy that is expressive and requires interpersonal processes which could be active or passive. In MI, a combination of the emotional, physical, social, mental, spiritual, and aesthetic aspects of music are used to maintain and improve the client's health condition. MI achieves its analgesic effects by acting on mu-opiate receptors, morphine-6-glucuronide and the level of interleukin-6. It could also compete with other peripheral nerve stimuli such as pain transmission to the brain via the spinal cord. MI also enacts a powerful and subtle psychological effect on people because it is rooted in their emotional lives. The psychological effect is rooted in the entrainment to the rhythm of the music which causes alteration of the neuron activities in the lateral temporal lobe.

A systematic review of literature conducted revealed that MI has been employed both in the preoperative phase for the management of anxiety and in the postoperative phase for the management of postoperative pain in breast cancer patients undergoing surgery. All the studies included in the systematic review used music that is culture-specific and face-to-face mode of delivery. None of the studies used theory-driven approach in their intervention development nor considered both preoperative and postoperative patient outcomes together.

Sequel to the recent global pandemic, many healthcare facilities are restricting access to patients in clinical settings creating limitations for music therapy interventions that rely on only face-to-face mode of delivery. Therefore, the delivery of music therapy via hybrid mode becomes an area worthy of research. As with the traditional delivery mode, the cultural context and the use of theory-driven intervention are considerations to be made when developing the intervention. In order to develop a theory-driven and culture-specific intervention, the Symptom Management Model (SMM) will be adopted in this study. SMM was selected based on the review of other literature on MI and considering the relatedness of components of MT and the components of the SMM.

Theoretical framework underpinning MI As stated previously, the SMM could underpin the MI in this study. The model was firstly developed by the School of Nursing symptom management faculty group of the University of California, San Francisco, and further revised. It has three domains which are symptom experience, symptom management strategy and symptom outcomes. The domains are dependent on the nursing concepts of person, environment, and health and illness. The symptom is described as a subjective experience that evinces a patient's biopsychosocial functioning, cognition, and sensation.

Symptom perception, evaluation and response to symptoms are the concepts indicated in the symptom experience domain. The symptom experience domain is directly influenced by risk factors or disease or injury and health status. For mastectomy patients, pain is usually influenced by the type of mastectomy and its extensiveness. However, the type of mastectomy to be done is dependent on the stage of cancer, the possibility of the patient undergoing radiotherapy, and the intended aesthetic result. The symptom management strategy domain is considered as a dynamic domain that aims at slowing down or averting negative outcomes using either professional, self-care, or biomedical strategies. MI is a type of intervention that can be used by both healthcare professionals and patients as an adjunct to pharmacological therapy for pain management. The components of the symptom management strategy include who delivers the intervention, what, how, when, why, where, and how much of the intervention is to be delivered. These are similar to the standards for reporting music intervention which includes consideration for the expertise, duration, frequency, dosage, mode of delivery and environment for the intervention to be delivered.

Finally, the symptom outcomes domain according to the SMM includes the effects of the intervention on the symptom status (pain intensity and analgesic consumption), functional status (vital signs), mood/emotional status (anxiety), and satisfaction with care. The SMM stresses that symptom experience assessment and adherence to the symptom management strategy will influence the outcomes achieved. Since pain is multidimensional, the amenability of each dimension to change by MI varies.

In relation to the findings that the cultural context in which MI will be implemented is crucial to the acceptance and effectiveness of the intervention and that symptom outcome in the SMM model in relation to MI for pain management can include symptom status (pain intensity and analgesic consumption), functional status (vital signs), mood/emotional states (anxiety), and satisfaction with care. To the best of our knowledge, an hybrid mode of delivering music intervention to women undergoing mastectomy has never been used to address postoperative pain. Given the strong relationship between music and pain, we hypothesize that the hybrid-mode delivered music therapy will reduce the preoperative anxiety, postoperative pain intensity, vital signs as well as improve satisfaction with pain management of women undergoing mastectomy. Therefore, this study aims to test the feasibility and evaluate the effectiveness of hybrid-mode delivered MI on preoperative anxiety, and acute postoperative pain, vital signs, analgesic consumption, and satisfaction with pain management among African women undergoing mastectomy.

Objectives of the study

The objectives of the study are to:

i) test the feasibility of implementing the MI intervention in clinical settings in Africa ii) Estimate the effects of MI on preoperative anxiety, acute postoperative pain, vital signs, analgesic consumption, and satisfaction with pain management among African women with breast cancer undergoing mastectomy

ELIGIBILITY:
Inclusion Criteria: Women who are:

1. Aged 18 years and above
2. Diagnosed with breast cancer
3. Attending the surgical out-patient clinic for booking visit
4. Being scheduled for mastectomy
5. Can communicate verbally or in writing in English, Yoruba or Pidgin;
6. Without existing chronic pain diagnosis
7. Consent to join the study. -

Exclusion Criteria:

1. Pre-existing mental health disorders and cognitive impairment if they are 2. Transferred to the intensive care unit due to complications within the first two days after surgery.

-

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women aged 18 and above diagnosed with breast cancer and undergoing mastectomy
Enrollment: 36 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-27 (Actual)

PRIMARY OUTCOMES:
Change in acute postoperative pain intensity | Pre-intervention and immediately after the intervention through study completion at 48 hours after surgery
  The Visual Analogue Scale will be used to assess the pain intensity level. The score on this scale ranged from 0 to 10, higher score represents high pain intensity

SECONDARY OUTCOMES:
Change in preoperative anxiety | Pre-intervention and immediately after the intervention on the day of surgery
  Spielberger State-Trait Anxiety Inventory will be used to assess anxiety level. This is a four point likert scale with score ranging from 0 to 80. Higher score represents high anxiety level.
Change in blood pressure | Pre-intervention and immediately after the intervention through study completion at 48 hours after surgery
  The systolic and diastolyic blood pressure will be assessed using an automated blood pressure monitor.
Analgesia consumption | Post-intervention at 48 hours after surgery
  The type, dosage, frequency and mode administration of analgesia will be assessed and documented in the pharmacological pain prescription and management technique chart.
Satisfaction with pain management | Immediately after intervention at 48 hours after surgery
  Patient satisfaction with pain management will be assessed using the numerical rating scale. The score on this scale ranged from 0 to 10, higher score represents high level of satisfaction
Change in heart rate | Pre-intervention and immediately after the intervention through study completion at 48 hours after surgery
  Heart rate will be assessed through an automated machine and documented in beats per minutes
Change in respiratory rate | Pre-intervention and immediately after the intervention through study completion at 48 hours after surgery
  Respiratory rate will be counted manually for one full minutes and documented as cycles per minute

CONTACTS AND LOCATIONS:
Overall Officials: Ka Ming Chow, DN, Study Chair — The Nethersole School of Nursing, Chinese University of Hong Kong
Locations (3):
- Kamuzu Central Hospital, Lilongwe, Malawi
- Nigeria (2):
  - Lagos State University Teaching Hospital, Ikeja, Lagos
  - Lagos University Teaching Hospital, Lagos

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to ensure privacy and confidentiality

REFERENCES:
- [Background] Anagnostopoulos, F., 2014. Mastectomy. Encycl. Qual. Life Well-Being Res. Well-Being Res. 141, 1077-1079. https://doi.org/10.1007/978-94-007-0753-5
- [Background] Andersen KG, Duriaud HM, Jensen HE, Kroman N, Kehlet H. Predictive factors for the development of persistent pain after breast cancer surgery. Pain. 2015 Dec;156(12):2413-2422. doi: 10.1097/j.pain.0000000000000298. PMID 26176893
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Binns-Turner PG, Wilson LL, Pryor ER, Boyd GL, Prickett CA. Perioperative music and its effects on anxiety, hemodynamics, and pain in women undergoing mastectomy. AANA J. 2011 Aug;79(4 Suppl):S21-7. PMID 22403963
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Cohen J. A power primer. Psychol Bull. 1992 Jul;112(1):155-9. doi: 10.1037//0033-2909.112.1.155. PMID 19565683
- [Background] Dion LJ, Engen DJ, Lemaine V, Lawson DK, Brock CG, Thomley BS, Cha SS, Sood A, Bauer BA, Wahner-Roedler DL. Massage therapy alone and in combination with meditation for breast cancer patients undergoing autologous tissue reconstruction: A randomized pilot study. Complement Ther Clin Pract. 2016 May;23:82-7. doi: 10.1016/j.ctcp.2015.04.005. Epub 2015 May 12. PMID 25986296
- [Background] Evans, H., 2019. Preoperative relaxation techniques for breast cancer patients undergoing breast-altering surgery: A systematic review. Iris J. Nurs. Care 1. https://doi.org/10.33552/ijnc.2019.01.000512
- [Background] Fecho K, Miller NR, Merritt SA, Klauber-Demore N, Hultman CS, Blau WS. Acute and persistent postoperative pain after breast surgery. Pain Med. 2009 May-Jun;10(4):708-15. doi: 10.1111/j.1526-4637.2009.00611.x. Epub 2009 Apr 22. PMID 19453965
- [Background] Fields LM, Calvert JD. Informed consent procedures with cognitively impaired patients: A review of ethics and best practices. Psychiatry Clin Neurosci. 2015 Aug;69(8):462-71. doi: 10.1111/pcn.12289. Epub 2015 Apr 13. PMID 25756740
- [Background] Gan TJ. Poorly controlled postoperative pain: prevalence, consequences, and prevention. J Pain Res. 2017 Sep 25;10:2287-2298. doi: 10.2147/JPR.S144066. eCollection 2017. PMID 29026331
- [Background] Gordon DB, Polomano RC, Pellino TA, Turk DC, McCracken LM, Sherwood G, Paice JA, Wallace MS, Strassels SA, Farrar JT. Revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R) for quality improvement of pain management in hospitalized adults: preliminary psychometric evaluation. J Pain. 2010 Nov;11(11):1172-86. doi: 10.1016/j.jpain.2010.02.012. Epub 2010 Apr 18. PMID 20400379
- [Background] Odejobi YO, Maneewat K, Chittithavorn V. Nurse-led post-thoracic surgery pain management programme: its outcomes in a Nigerian Hospital. Int Nurs Rev. 2019 Sep;66(3):434-441. doi: 10.1111/inr.12515. Epub 2019 Jul 19. PMID 31322292